CLINICAL TRIAL: NCT05944796
Title: Diathermy Effectiveness in Reducing Subcutaneous Adipose Tissue Affected by Lipedema
Acronym: EDRTASAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Principal Investigator, Edurne Úbeda D'Ocasar, Doctor Edurne Úbeda D'Ocasar, Camilo Jose Cela University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CamiloJcUDL
Record Dates: First submitted 2023-06-19; First posted 2023-07-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lipedema
Keywords: Lipedema
MeSH Terms: conditions — Lipedema | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diathermy (Experimental): The experimental group will receive 10 diathermy sessions.
  Interventions: Other: Diathermy
- Placebo (Placebo Comparator): The placebo comparator, will receive 10 placebo sessions.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Diathermy — The patients belonging to the experimental group will undergo 10 diathermy sessions. The control group will have the same sessions but in athermy (placebo)
  Arms: Diathermy
Other: Placebo — The patients belonging to the placebo group will undergo 10 placebo sessions (athermya)
  Arms: Placebo

SUMMARY:
Diathermy, a therapy that uses deep heat to reach deep tissue layers, is known to induce the breaking down of fatty cells and fibrotic tissue. In lipedema, patients develop fibrosis of their subcutaneous adipose tissue. Therefore, diathermy could be an interesting tool to treat this disease. To test the effectiveness of diathermy on these patients, the investigators will select women with lipedema (18 to 70 yo) and place them in two groups (experimental and control group). The experimental group will receive the treatment, that is, 10 minutes of diathermy on the medial knee surface of both knees, with an intensity that produces heat just below the participants' pain threshold. Participants from the control group will receive sham diathermy, that is, placebo. The intervention consists of 10 sessions, 3 times a week, for 4 weeks. Researchers will collect data pre and post intervention and one month after the intervention ends. Data will consist of measurements at knee level with tape and an ultrasound device, pain threshold with an algometer, a VAS score and an SF-12 questionnaire for quality of life.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test the effectiveness of diathermy in reducing the subcutaneous adipose tissue affected by lipedema in women suffering from this disorder. The main questions it aims to answer are:

* Does diathermy produce changes in subcutaneous adipose tissue affected by lipedema?
* Is it effective as a tool for lipolysis and/or fibrolysis of said subcutaneous adipose tissue affected by lipedema?
* Do these changes result in a reduction of subcutaneous adipose tissue affected by lipedema?
* Do these changes decrease pain in the area treated with diathermy?

Participants will:

* Be assesed prior to receiving treatment:

  * Circometry of both knees (at joint space level)
  * Pain threshold using an algometer. Area: medial below knee region, at fibular head level
  * SF-12 questionnaire
  * VAS score
  * Ultrasound mesurements at medial collateral ligament (distance from skin to ligament)
* Receive 10 diathermy sessions. 10 minutes per knee (medial knee surface), 3 times a week for 4 weeks. Parameters: 470 KHz, capacitive head, intensity: heat below pain threshold.
* Be assesed after receiving treatment:

  * Circometry of both knees (at joint space level)
  * Pain threshold using an algometer. Area: medial below knee region, at fibular head level
  * SF-12 questionnaire
  * VAS score
  * Ultrasound mesurements at medial collateral ligament (distance from skin to ligament)
* Be assesed after receiving treatment (one month post intervention):

  * Circometry of both knees (at joint space level)
  * Pain threshold using an algometer. Area: medial below knee region, at fibular head level
  * SF-12 questionnaire
  * VAS score
  * Ultrasound mesurements at medial collateral ligament (distance from skin to ligament)

Researchers will compare an experimental group to a placebo group to see if treatment with diathermy is effective in reducing subcutaneous adipose tissue affected by lipedema.

ELIGIBILITY:
Inclusion Criteria:

* women between 18-70 years old.
* Diagnosed with lipedema by a medical service.
* Patients with type III or V lipedema (involvement of legs).
* Patients with type II lipedema are also admitted if they have a fat pad on the inner side of the knee

Exclusion Criteria:

* Pregnant
* Pacemaker or some other electronic implant
* Metal implants or knee prostheses
* Open wounds or burns on the inside of the knee
* Thrombophlebitis
* Malignant growths (cancer)
* Infectious processes
* Follow other non-conservative treatment related to lipedema at that time

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change of adipose tissue in the knee | baseline
  Using ultrasound, it is intended to know if a reduction in adipose tissue has occurred after the application of diathermy.
Change of adipose tissue in the knee | after finishing the treatment (one month)
  Using ultrasound, it is intended to know if a reduction in adipose tissue has occurred after the application of diathermy.
Change of adipose tissue in the knee | 30 days after finishing the treatment.
  Using ultrasound, it is intended to know if a reduction in adipose tissue has occurred after the application of diathermy.
Contour change in the knee. | baseline
  By using a tape measure, the circummetry of the knees on both sides will be assessed. The greater the contour, the more volume the patient will show.
Contour change in the knee. | after finishing the treatment (one month)
  By using a tape measure, the circummetry of the knees on both sides will be assessed. The greater the contour, the more volume the patient will show.
Contour change in the knee. | 30 days after finishing the treatment.
  By using a tape measure, the circummetry of the knees on both sides will be assessed. The greater the contour, the more volume the patient will show.
Quality of life (SF-12). | baseline
  SF-12 quality of life questionnaire. The higher the score obtained in the questionnaire, the better the patient's quality of life. The maximum value that can be reached is 100 and the minimum is 0.
Quality of life (SF-12). | after finishing the treatment (one month)
  SF-12 quality of life questionnaire. The higher the score obtained in the questionnaire, the better the patient's quality of life. The maximum value that can be reached is 100 and the minimum is 0.
Quality of life (SF-12). | 30 days after finishing the treatment.
  SF-12 quality of life questionnaire. The higher the score obtained in the questionnaire, the better the patient's quality of life. The maximum value that can be reached is 100 and the minimum is 0.
Measure pain | baseline
  Visual analogic scale (VAS). The higher the visual analogue scale score, the more pain the patient presents. The maximum value that can be reached is 10 and the minimum is 0.
Measure pain | after finishing the treatment (one month)
  Visual analogic scale (VAS). The higher the visual analogue scale score, the more pain the patient presents. The maximum value that can be reached is 10 and the minimum is 0.
Measure pain | 30 days after finishing the treatment.
  Visual analogic scale (VAS). The higher the visual analogue scale score, the more pain the patient presents. The maximum value that can be reached is 10 and the minimum is 0.
Algometry. | baseline
  Using the algometer, pain sensitivity will be assessed when pressing medial infracondylar leg at the level of the fibular head. The lower the algometry score, the more pain the patient will have. The maximum value that can be reached is 5 and the minimum value is 0.
Algometry. | after finishing the treatment (one month)
  Using the algometer, pain sensitivity will be assessed when pressing medial infracondylar leg at the level of the fibular head. The lower the algometry score, the more pain the patient will have. The maximum value that can be reached is 5 and the minimum value is 0.
Algometry. | 30 days after finishing the treatment.
  Using the algometer, pain sensitivity will be assessed when pressing medial infracondylar leg at the level of the fibular head. The lower the algometry score, the more pain the patient will have. The maximum value that can be reached is 5 and the minimum value is 0.

SECONDARY OUTCOMES:
Sociodemographic variables | baseline.
  Sociodemographic data such as age, weight, height and marital status will be collected

CONTACTS AND LOCATIONS:
Locations (1):
- University Camilo José Cela, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No